CLINICAL TRIAL: NCT05824624
Title: The Effect Of Animal-Assisted Intervention On Fear In Hospıtalızed Children In The Emergency Department: A Randomized Controlled Study
Brief Title: The Effect Of Animal-Assisted Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mukaddes Demir Acar, Ass. Prof., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DEMIRACAR
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Animal Model; Pediatric; Emergencies; Fear; Nursing Caries
MeSH Terms: conditions — Disease Models, Animal; Emergencies

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental model
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Animal-supported application will be made to the children in the study group.
  Interventions: Other: ANIMAL-ASSISTED INTERVENTION
- control group (Experimental): Routine care will be given to the children in the control group.
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: ANIMAL-ASSISTED INTERVENTION — It will be ensured that the child is introduced to the goldfish when he is lying in the observation room, that the child will name the fish, and that he will communicate and feed the fish during his stay. Thus, it is aimed to turn the attention of the child to the goldfish while in the emergency room, to distract the child with the fish while all nursing interventions are presented, and to reduce the fear.
  Arms: study group
Other: Routine Care — Routine nursing care will be provided.
  Arms: control group

SUMMARY:
The aim of the study is to examine the effect of animal-assisted practice on fear in children admitted to the emergency room.

DETAILED DESCRIPTION:
Children's fears about the hospital are traumatic and confront us as a hindering factor in their growth and development.Bringing the child to the emergency room and not knowing what will happen there creates great fear in him. Children already have different fears according to different age groups and developmental stages. These; separation from family, pain and suffering, change in body image (losing body parts), etc. The state of fear can lead to a worsening of the child's existing illness and symptoms. In addition to being separated from the family, being separated from peers, not being able to play games, staying away from school if going to school, etc. they have concerns.

ELIGIBILITY:
Inclusion Criteria:

* To be followed for at least 2 hours in the pediatric emergency room,
* Age range is 5-7,
* Not afraid of the goldfish to be used in the research,
* Not allergic to fish and fish feed,
* Does not have physical, auditory, visual and cognitive barriers to feeding (feeding),
* No speech or communication disorder that will prevent the parent and child from communicating,
* Parent and child's willingness to participate in the research

Exclusion Criteria:

* Patients who are not admitted to the Pediatric Emergency room, patients who do not fit the age range of 5-7, who stay less than 2 hours,
* Afraid of goldfish, allergic to fish food, preventing feeding, having physical, auditory, visual and cognitive disabilities,
* Patients with speech and communication disorders that will prevent parents and children from communicating,
* Parent and child not willing to participate in the research.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
The Scale Development of Fear in Children Against Nursing Interventions and Used Materıals | 2 hours
  The scale was created to develop a valid and reliable measurement tool for children to determine their fear of nursing interventions and used materials. As a result of the validity and reliability analyzes of the scale, it was composed of 18 items. The scale has 2 sub-dimensions. These are fear of common materials (10 items) and fear of uncommon materials (8 items). The scale was scored as (1) not afraid, (2) little afraid, (3) afraid, (4) very afraid, (5) extremely afraid.
Child Fear Scale | 2 hours
  The Scale is a scale consisting of the display of five drawn facial expressions, ranging from neutral expression (0 points) to "no fear" to frightened face (4 points) to "severe fear". The scale is intended for children aged 5-10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mukaddes Demir Acar, Principal Investigator — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Özalp Gerçeker, G., Ayar, D., Özdemir, Z., & Bektaş, M. 2018. Gaining of Children's State Anxiety and Children's Fear Scale to Turkish Language. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 11(1), 9-13.
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Result] Eren Kok H, Orsal O. The Development of a Scale to Measure Children's Fear of Nursing Interventions and Instruments Used in Hospital. Psychiatry and Behavioral Sciences 2023;13(1):47-56. Doi: 10.5455/PBS.20221101060619